CLINICAL TRIAL: NCT00659204
Title: A Randomized Controlled Trial of the Efficacy of a Novel Silver Nanoparticle Gel Versus a Common Antibacterial Hand Gel Against Bacterial Hand Flora
Brief Title: Efficacy of Silver Nanoparticle Gel Versus a Common Antibacterial Hand Gel
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Researcher left the institution
Sponsor: Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 208035
Record Dates: First submitted 2008-04-11; First posted 2008-04-16 (Estimated); Results first posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Silver Nanoparticle Gel (Experimental): Silver Nanoparticle Gel (SilvaSorb, AcryMed, Inc., Portland, OR)
  Interventions: Drug: Silver Nanoparticle Gel
- alcohol-based gel (Active Comparator): Alcohol-based hand gel (Purell, GoJo Industries, Akron, OH)
  Interventions: Drug: alcohol-based hand gel

INTERVENTIONS:
Drug: Silver Nanoparticle Gel — SilvaSorb® gel applied topically to the hands with a limited exposure time of 10 minutes
  Other Names: SilvaSorb® gel
  Arms: Silver Nanoparticle Gel
Drug: alcohol-based hand gel — Purell gel applied topically to the hands with a limited exposure time of 10 minutes
  Other Names: Purell
  Arms: alcohol-based gel

SUMMARY:
The purpose of this pilot study is to compare the antimicrobial efficacy of silver nanoparticle gel to a commercialized alcohol-based hand gel on bacterial counts isolated from the hands of 40 volunteers seeded with Serratia marcescens, a surrogate microbial marker. Specific aims of this study are: Aim #1: Compare the immediate antimicrobial efficacy of a one-time application of silver nanoparticle gel (SilvaSorb , AcryMed, Inc., Portland, OR) versus an alcohol-based hand gel (Purell, GoJo Industries, Akron, OH) in reducing transient bacterial counts isolated from hands seeded with S. marcescens.

Aim # 2: Compare the persistent antimicrobial efficacy of a one-time application of silver nanoparticle gel (SilvaSorb) versus an alcohol-based hand gel (Purell) over a 10 minute time frame in producing a persistent reduction on transient bacterial counts isolated from hands seeded with S. marcescens.

Aim # 3: Compare user acceptability of silver nanoparticle gel (SilvaSorb) versus an alcohol-based hand gel (Purell) using a self-assessment questionnaire.

DETAILED DESCRIPTION:
The objective of this randomized controlled, double blinded, 2x3 experimental study is to evaluate the antimicrobial efficacy of silver nanoparticle gel compared to an alcohol-based hand gel on bacterial counts isolated from the hands of 40 healthy, adult, military student volunteers. The study will be conducted in two phases: the first phase will consist of a methods development period and the second phase will consist of the formal pilot study. For phase I, the first four participants from the sample pool will be assigned into one of two groups (nano-silver gel or alcohol-based gel) whereas in Phase II, the participants will be randomized into one of two groups. Participants in both phases will follow a 7 day washout period where subjects will refrain from using antimicrobial products for a week prior to testing. Testing of participants in both phases will start with a baseline bacterial hand count. This will be accomplished by using a surrogate biomarker (S. Marcescens). This microorganism was selected because it is considered the standard surrogate marker to be used in hand hygiene evaluations and because it produces a characteristic red colony that is easily distinguishable from normal microbial populations of the hands making colony counting more accurate. Sampling of bacterial flora will be accomplished utilizing an established "modified glove juice" technique in which the participant's dominant hand is placed into a large sterile bag containing a sampling solution, which removes the surrogate bacteria. Once baseline samples have been collected, all participants will then complete two additional random ordered timed conditions involving the surrogate biomarker and one of the two test gels. For each test condition, five mL of solution will be withdrawn from the collection bag, diluted, plated, and incubated for 36 hours. For the immediate efficacy testing, a glove juice sampling will be obtained after a 1 minute application of the gel. For the persistent efficacy testing, a glove juice sampling will be obtained after a 10 minute application of the gel. To ensure the biomarker has been removed, all subjects will wash hands with a 70% ethanol surgical handwash. The use of an UV-C light will also be implemented for 20 seconds as an additional precaution. Participants in phase I will have an additional glove juice sampling at the end of degerming to validate the protocol. All participants will end the study by completing a 4 question visual analog questionnaire to determine user acceptability of the gels. The percent difference of total bacterial counts from baseline will be used as the outcome variable. An unpaired Student's t-test (or an appropriate non-parametric test) will be used for data analysis for each of the study aims.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Ability to read and understand English (for consent purposes)
* Free of clinically evident dermatitis, open wounds, sores, or breaks in hand skin determined by a Visual Skin Scale (VSS).
* Free of hand jewelry or artificial nail enhancements
* Have fingernails that are clean and extend no longer than approximately one (1) mm past the nail bed

Exclusion Criteria:

* Anyone directly working in a healthcare, public health, or long term residence setting.
* Currently receiving any antibiotics, or on any other in as investigational drug, steroids or immunosuppressive therapy.
* Reports cuts, scratches, or skin disorders, or Dermatitis visualized by the PI/AI using the Visual Skin Scale (VSS).
* Reports any form of current immune disorders such as AIDS, lupus, any cancers (solid or hematopoietic), or other medical conditions such as diabetes, hepatitis, rheumatoid arthritis, or an organ transplant recipient.
* Known sensitivities or allergies to silver, alcohol, latex, soap, detergent, antibiotics.
* Any use of artificial nail enhancements or any non-removable rings
* Primary care provider or resident in a setting where someone has known impaired immunocompetence (currently receiving chemotherapy, HIV positive), requires wound care or intravenous management.
* Currently pregnant/lactating or taking care of children under the age of 3 or anyone that requires diaper changing.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary S McCarthy, PhD, MN, Principal Investigator — Nurse Scientist, Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center, Tacoma, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We assessed 24 subjects for eligibility. 2 did not meet inclusion criteria which left us with 22 subjects who were randomized into two groups; 11 in each group.
Groups:
- Nano-silver Gel: Silver Nanoparticle Gel (SilvaSorb, AcryMed, Inc., Portland, OR)
Period: Overall Study
Arm/Group | Nano-silver Gel | Alcohol-based Gel
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nano-silver Gel | Alcohol-based Gel | Total
Number analyzed (Participants) | 11 | 11 | 44
Age, Categorical [Count of Participants; unit: Participants]
  number analyzed (Participants) | 11 | 11 | 22
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: particpants]
  Female: number analyzed (Participants) | 11 | 11 | 22
  Female | 0 | 0 | 0
  Male: number analyzed (Participants) | 11 | 11 | 22
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  United States: number analyzed (Participants) | 11 | 11 | 22
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Microbial Count at Baseline
Description: Subjects' hands are contaminated with 1.5 milliliters (mL) aliquot of S. marcescens which is then distributed evenly over both hands. A 30 second massage with bacteria followed by one minute of timed air drying takes place prior to the modified glove juice sampling procedure. Subject's dominant hand is placed into a sterile 1 liter polyethylene bag with 75 mL of sampling solution. Hand is removed after 60 seconds of massage and 5 mL of juice is retrieved, diluted 1:10 within 5 minutes, and plated in duplicate on trypticase soy agar. Samples are transported in bio-transport container to the lab where they are incubated aerobically at 36 degrees Centigrade for 36 hours.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Nano-silver Gel | Alcohol-based Gel
Number analyzed (Participants) | 11 | 11
CFU/mL | 105 (7.1) | 107 (8.1)

2. Secondary Outcome: User Acceptability
Description: User Acceptability Questionnaire - Self-assessment. Investigator-developed instrument that included 4 questions regarding the specific hand gel product applied to the participant's hands: 1) I would rate my acceptance of this product as?; 2) I would consider using this product again?; 3) I would rate my confidence in this product as?; and 4) I would recommend using this product to my co-workers?. Scale had anchors of 1 (least acceptable) to 10 (most acceptable). Total score was the sum of scores for each of the 4 questions; range was 4 to 40. there were no subscales. A score of 4 demonstrated least acceptance and score of 40 demonstrated highest acceptance.
Time Frame: 2 hours
Population: Data from all participants could be used, there were no dropouts.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nano-silver Gel | Alcohol-based Gel
Number analyzed (Participants) | 11 | 11
score on a scale | 27 (5.7) | 33 (5.6)

3. Primary Outcome: Microbial Count - Persistent Effect
Description: Microbial count of hands seeded with S. marcescens after ten minutes of exposure and treatment with an antimicrobial gel. Same modified glove juice sampling technique was used and 1.5 milliliters of juice was removed, diluted, and plated for incubation.
Time Frame: 10 minutes
Population: Everyone was included, there were no drop outs.
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Nano-silver Gel | Alcohol-based Gel
Number analyzed (Participants) | 11 | 11
CFU/mL | 65 (9.4) | 103 (8.7)

4. Primary Outcome: Microbial Count - Immediate Effect
Description: Subjects underwent the modified glove juice technique after seeding of hands with S. marcescens bacteria for 1 minute followed by application of one of the two antimicrobial gels; a 1.5 milliliter sample of the juice was collected after 1 minute. The procedure was repeated for each of the two gels, random order assigned.
Time Frame: 1 minute
Population: All subjects included, there were no drop outs.
Measure: Mean (Standard Deviation); unit: CFU/mL
Arm/Group | Nano-silver Gel | Alcohol-based Gel
Number analyzed (Participants) | 11 | 11
CFU/mL | 101 (6.6) | 49 (10.2)

ADVERSE EVENTS:
Time Frame: 48 hours
Description: The intervention took place on one day only. We followed up with subjects for potential adverse events in the subsequent 24 hours for a total of 48 hours.
Arm/Group | Nano-silver Gel | Alcohol-based Gel
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
Further investigation is warranted to test silver nanoparticle gel as a persistent antibacterial therapeutic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No